CLINICAL TRIAL: NCT05112016
Title: Long-term Cohort Study of Mesorectal Excision for Rectal Cancer
Acronym: TME-KSW
Status: Recruiting | Type: Observational
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Other Study IDs: TME-KSW
Record Dates: First submitted 2021-09-06; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-09

CONDITIONS: Rectum; Cancer
Keywords: TME (total mesorectal excision); Transanal TME; Laparoscopic TME; Robotic TME; Open TME; Quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TME for rectal cancer: Patients with rectal cancer treated by TME (laparoscopic TME, transanal TME, robotic TME, open TME)
  Interventions: Procedure: Total mesorectal excision for rectal cancer

INTERVENTIONS:
Procedure: Total mesorectal excision for rectal cancer
  Other Names: TME

SUMMARY:
The aim of this cohort study is to record, evaluate and compare the surgical, oncological as well as the functional outcome and Quality of life after mesorectal excision for rectal cancer

DETAILED DESCRIPTION:
Outcomes of mesorectal excision patients will be analysed. Medical records will be reviewed and perioperative outcomes retrieved, incl. long-term oncological and functional/quality of life data. A retrospective cohort over 10 years (2007-2016) will serve as a control to a prospective cohort over 10 further years (2017-2026) as to investigate trends in perioperative and oncological outcomes (min. follow-up of 5 years + adequate cohort size). Prospective data on bowel function, urogenital function and quality of life will measured at time of diagnosis and further. Variations in neoadjuvant/adjuvant treatment and surgical approaches will be assessed for their effect on the outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women >18 years
* Patients with rectal cancer
* Underwent mesorectal excision
* Agreed to fill in a validated questionnaires before surgery and after stoma reversal
* Informed consent

Exclusion Criteria:

* Age < 18
* No informed consent (no general consent, no consent to use personal data for research purpose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rectal cancer who benefit from surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative mortality | 90 days
  Reporting perioperative mortality with Clavien-Dindo & Comprehensive Complications Index
Age | 10 years
  Age (years)
Body mass index | 10 years
  BM (kg/m2)
Gender | 10 years
  Sex (male, female)
ASA score | 10 years
  American Society of Anesthesiologists score (I to V)
Date of surgery | day of surgery
  date of surgery (day-month-year)
Tumor localisation | 10 years
  Description of tumor localisation
Comorbidities | day of surgery
  Charlson index
Perioperative complications | 90 days
  Reporting and grading of postoperative surgical complications (according to Dindo-Clavien classification and/or comprehensive complications index)
Histological results | 30 days
  Histological staging and grading of the specimen by a pathologist
Quality of life, including functional and symptom scales, incontinence scores, sexual function | 10 years
  taTME survey (validated english, german, french versions); from 0 (worst) to 100 (best)

SECONDARY OUTCOMES:
Perioperative treatment | 10 years
  Chemoradiation before or after surgery, other treatments necessary
Surgery time | day of surgery
  Duration of surgery in minutes
Length of hospital stay | 90 days
  Length of hospital stay in days
Readmission rate | 90 days
  Number of patients readmitted within 90 days of index surgery divided by the total number of patients operated
Costs | 10 years
  At the level of individual patient Cost in terms of hospital charges and expenses in Swiss Francs. Actual costs and micro-costing

CONTACTS AND LOCATIONS:
Overall Officials: Michel Adamina, Prof/MD/MSc, Principal Investigator — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided